CLINICAL TRIAL: NCT02429037
Title: Recombinant Adenoviral Human p53 Gene Combined With Radio- and Chemo-therapy in Treatment of Unresectable, Locally Advanced Head and Neck Cancer - a Open-labeled Randomized Phase 2 Study
Brief Title: P53 Gene Combined With Radio- and Chemo-therapy in Treatment of Unresectable Locally Advanced Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen SiBiono GeneTech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rAd-p53-J1002
Record Dates: First submitted 2015-04-20; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-03

CONDITIONS: Advanced Head and Neck Cancer
Keywords: p53; gene therapy; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiation; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rAd-p53 plus radiation and chemotherapy (Experimental): rAd-p53 tumor injection combined with radio- and chemo-therapy.
  Interventions: Drug: rAd-p53; Radiation: radiation; Drug: Cisplatin
- radiation and chemotherapy (Active Comparator): radiation combined with chemotherapy
  Interventions: Radiation: radiation; Drug: Cisplatin

INTERVENTIONS:
Drug: rAd-p53 — multi-point injections of rAd-p53 into tumor on day 1, 8 and 15 at a dose of 2 × 10^12 viral particles (VP) in a 21-days cycle.
  Other Names: p53 gene therapy
  Arms: rAd-p53 plus radiation and chemotherapy
Radiation: radiation — radiation therapy will be given at a total dose of 60 Gy by 2.0 Gy/fraction, daily Monday-Friday for 6 weeks.
Drug: Cisplatin — Cisplatin 100 mg/m2 IV on days 1 plus paclitaxel 30 mg/m2 IV on day 1, 8 and 15
  Other Names: chemotherapy: cisplatin

SUMMARY:
The objectives of this study are to investigate the efficacy and safety of rAd-p53 gene combined with radio- and chemo-therapy vs. radio- and chemo- therapy only in treatment of unresectable, locally advanced head and neck cancer. This is a phase 2, open labeled, and active-controlled study.

DETAILED DESCRIPTION:
To evaluate benefits of rAd-p53) gene therapy combined with radio- and chemo-therapy in treatment of unresectable, locally advanced head and neck cancer, total of 60 patients with above condition will be randomly assigned to two groups: the experiment group (EG) and the control group (CG). The EG received multi-point injections of rAd-p53 into tumor on day 1, 8 and 15 at a dose of 2 × 10^12 viral particles (VP) in a 21-days cycle. Both EG and CG were given radiotherapy at a total dose of 60 Gy and chemotherapy (Cisplatin 100 mg/m2 IV on days 1 plus paclitaxel 30 mg/m2 IV on day 1, 8 and 15). The patients will be treated until disease progression, withdrawal from study, or untolerated adverse events. study endpoints are efficacy (Progression-free survival, overall survival) and safety variables.

ELIGIBILITY:
Inclusion Criteria:

1. histopathologically diagnosed head and neck cancer;
2. unresectable, locally advanced;
3. 18 years or older;
4. with an Eastern Cooperative Oncology Group (ECOG) score of 0-2;
5. with normal tests of hemogram, blood coagulation, liver and kidney function; 6.signed the informed consent form.

Exclusion Criteria:

1. Serious blood coagulation disorder, bleeding tendency, platelet < 6 * 1000000000/L;
2. have serious heart, lung function abnormalities or severe diabetes patients;
3. active infection;
4. severe atherosclerosis;
5. AIDS patients;
6. serious thrombotic or embolic events within 6 months;
7. renal insufficiency requiring hemodialysis or peritoneal dialysis;
8. pregnant or lactating women;
9. mental disorder or disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | three years after starting treatment
  Patients will be followed up until progression or death, withdrawal from study, or until data cut-off after 3 years.

SECONDARY OUTCOMES:
Adverse events | from starting study treatment until 30 days after the last study treatment
  Adverse events
overall survival | three years after starting study treatment
  Patients will be followed up until death, withdrawal from study, or until data cut-off after 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu cancer hospital, Nanjing, Jiangsu, China